CLINICAL TRIAL: NCT01880125
Title: Clinical Trial to Compare the Pharmacokinetics Profile of YJAT Sustained Release Tablet and ULTRACET® Immediate Release Tablet After Oral Administration to Healthy Male Subjects
Brief Title: Assessment of the Pharmacokinetics of a Sustained Release Formulation of a Tramadol/Acetaminophen Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Collaborators: Chonbuk National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: YJ4-101
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Pain
Keywords: Tramadol; Acetaminophen; Pharmacokinetics; Sustained release; Immediate release
MeSH Terms: conditions — Pain | interventions — Ultracet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): Period 1: Tramadol HCI/Acetaminophen 37.5/325mg PO once with water 240ml at fasted state Period 2: Tramadol HCI/Acetaminophen 75/650mg PO once once with water 240ml at fasted state
  Interventions: Drug: Tramadol HCI/Acetaminophen
- Group B (Other): Period 1: Tramadol HCI/Acetaminophen 75/650mg PO once once with water 240ml at fasted state Period 2: Tramadol HCI/Acetaminophen 37.5/325mg PO once with water 240ml at fasted state
  Interventions: Drug: Tramadol HCI/Acetaminophen

INTERVENTIONS:
Drug: Tramadol HCI/Acetaminophen — Test drug: Tramadol HCI/Acetaminophen 75/650mg, two times daily. Reference drug: Tramadol HCI/Acetaminophen 37.5/325 mg, four times daily.
  Other Names: ULTRACET immediate release tablet; YJAT sustained release tablet

SUMMARY:
1. Objective: To evaluate the pharmacokinetic profiles of an SR 75 mg tramadol/650 mg acetaminophen formulation compared with an immediate release (IR) 37.5 mg tramadol/325 mg acetaminophen formulation after a single dose and at steady state
2. Subjects: Healthy subject
3. Methods: A phase I study to evaluate the pharmacokinetic sustained release and immediate release treatment profiles at steady state.

DETAILED DESCRIPTION:
This study was open, randomized, 2-period, 2-treatment multiple-dose crossover study of immediate release treatment and sustained release treatment was designed to assess the pharmacokinetics after a 2-day repeated administration in which the steady state was achieved.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 20 and 45 years
* Subjects weighed ≥ 45 kg and were within 20% of their ideal body weight
* No clinically relevant abnormalities identified by vital sign measurement, 12-lead electrocardiography and routine laboratory test

Exclusion Criteria:

* Hypersensitivity or histories of sensitivity to either tramadol or acetaminophen
* Evidence or histories of clinically significant renal, digestive, respiratory, musculoskeletal, endocrine, psychiatric, neurological, hematological or cardiovascular diseases
* Taking any prescription or herbal medicines within 2 weeks before the study or any over-the-counter medication within 1 week before the study
* Systolic blood pressure (SBP) ≥ 160 mmHg or ≤ 100 mmHg or diastolic blood pressure (DBP) ≥ 95 mmHg or ≤ 60 mmHg
* Any surgical or medical conditions that could affect drug absorption

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetic profiles of tramadol and acetaminophen at steady state | 0 to 36 hour
  Bio-equivalence of Cmax at steady state of tramadol and acetaminophen
Evaluate the pharmacokinetic profiles of tramadol and acetaminophen at steady state | 0 to 36 hour
  Bio-equivalence of AUC at steady state of tramadol and acetaminophen

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics profiles of tramadol, acetaminophen and O-desmethyltramadol at steady state | 0 to 36 hour
  Tmax of tramadol and acetaminophen at steady state.
Evaluate the pharmacokinetics profiles of tramadol, acetaminophen and O-desmethyltramadol at steady state | 0 to 36 hour
  Half-life of tramadol and acetaminophen at steady state.
Evaluate the pharmacokinetics profiles of tramadol, acetaminophen and O-desmethyltramadol at steady state | 0 to 36 hour
  Accumulation index of tramadol and acetaminophen at steady state.
Evaluate the pharmacokinetics profiles of tramadol, acetaminophen and O-desmethyltramadol at steady state | 0 to 36 hour
  Cmax of O-desmethyltramadol at steady state
Evaluate the pharmacokinetics profiles of tramadol, acetaminophen and O-desmethyltramadol at steady state | 0 to 36 hour
  AUC of O-desmethyltramadol at steady state
Evaluate the pharmacokinetics profiles of tramadol, acetaminophen and O-desmethyltramadol at steady state | 0 to 36 hour
  Tmax of O-desmethyltramadol at steady state
Evaluate the pharmacokinetics profiles of tramadol, acetaminophen and O-desmethyltramadol at steady state | 0 to 36 hour
  Half-life of O-desmethyltramadol at steady state

REFERENCES:
- [Derived] Im YJ, Jeon JY, Kim EY, Kim Y, Oh DJ, Yoo JS, Shin DH, Chae SW, Kim MG. An assessment of the pharmacokinetics of a sustained-release formulation of a tramadol/acetaminophen combination in healthy subjects. Clin Ther. 2015 Feb 1;37(2):376-89. doi: 10.1016/j.clinthera.2014.12.007. Epub 2015 Jan 22. PMID 25618318